CLINICAL TRIAL: NCT06992102
Title: Clinical Study on the Treatment of Lower Respiratory Tract Infection With Pseudomonas Aeruginosa by Ceftazidime and Avibatam
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-SR-500
Record Dates: First submitted 2025-04-17; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: MDRPA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multidrug-resistant Gram-negative bacteria (MDR-GNB) is emerging globally as a pathogen of concern in healthcare-associated infections (HAIs), and a threat to public health.There has been an alarming rise in the prevalence of MDR-GNB infections globally over the last decade.Multidrug-resistant or Carbapenem-resistant Pseudomonas aeruginosa (MDRPA or CRPA) are one of the major pathogens in the hospital setting,and are particularly challenging due to limited therapeutic options,associated with high mortality rates.Ceftazidime/avibactam(CAZ/AVI) combines the anti-pseudomonal cephalosporin ceftazidime and the novel non-β-lactam β-lactamase inhibitor avibactam,which are now available for the treatment of MDR-GNB infections and favorable outcomes have been reported in hospitalized patients with carbapenem-resistant Enterobacterales (CRE).However, there are only few publications available with a small sample size limit, focusing on the efficacy of CAZ/AVI for the treatment of CRPA or MDRPA infections.Therefore, a retrospective analysis was conducted to compare the clinical efficacy and microbiological efficacy of CAZ/AVI versus other antibiotics for the treatment of MDRPA infections.

ELIGIBILITY:
Inclusion Criteria:

* patients with MDRPA infection diagnosed by clinicians
* patients treated with anti-Pseudomonas aeruginosa antibiotics for at least 72h
* patients older than 18 years old.

Exclusion Criteria:

* Patients with human immunodeficiency virus infection, mental illness, a medication course of less than 72 hours, or incomplete data were excluded.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This was a single-centre, retrospective and observational study conducted in the First Affiliated Hospital of Nanjing Medical University, a 2200-bed tertiary care teaching hospital in Nanjing, Jiangsu in China, from January 2019 to April 2023.The inclusion criteria consisted of (i) patients with MDRPA infection diagnosed by clinicians,(ii) patients treated with anti-Pseudomonas aeruginosa antibiotics for at least 72h,(iii) patients older than 18 years old. Patients with human immunodeficiency virus infection, mental illness, a medication course of less than 72 hours, or incomplete data were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy | 28 day after enrollment
  The clinical efficacy of the treatment was determined by two senior physicians with extensive clinical experience, who classified it as either effective (characterized by the resolution or significant improvement of clinical symptoms and signs, normalization or minimal residuals in pulmonary imaging, and normalization of inflammatory markers), uncertain or ineffective.

SECONDARY OUTCOMES:
Microbiological efficacy | 28 day after enrollment
  Microbiological efficacy was defined as eradication or reduction, indicated by the absence of MDRPA in lower respiratory tract secretion cultures post-treatment, or a decrease in bacterial load by more than 25% compared to pre-treatment levels. Microbiological ineffectiveness was defined as the continued presence of MDRAB in cultures after treatment and no change or an increase in bacterial load compared to pre-treatment levels.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China